CLINICAL TRIAL: NCT03605043
Title: Integrated Hypertension and HIV Care Cascades in a HIV Treatment Program in Eastern Uganda: a Retrospective Cohort Study
Brief Title: Integrated Hypertension and HIV Care Cascades in Uganda
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: ss 4583
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Hypertension; HIV
Keywords: Integrated; Care cascade; Uganda
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall cohort: All Persons Living with HIV who enlisted in any one of three high-volume HIV clinics in Tororo District of Eastern Uganda between 2014 and 2017.
  Interventions: Other: Blood pressure management in the HIV program

INTERVENTIONS:
Other: Blood pressure management in the HIV program — Integrated care for hypertension and HIV in the HIV program

SUMMARY:
In this retrospective cohort study, we mapped the care cascades for both Hypertension and HIV within a HIV program in Uganda with the goal of identifying opportunities for developing contextually appropriate integrated care models, .

DETAILED DESCRIPTION:
Persons living with HIV (PLHIV) and receiving anti-retroviral therapy (ART) are at increased risk of cardiovascular disease (CVD) due to direct effects of ART and HIV infection itself, compounded by traditional CVD risk factors such as increased life expectancy and Westernized diet. Additionally, in sub-Saharan Africa, as is the case globally, hypertension (HTN) is a major risk factor for CVD. The prevalence of HTN in the setting of HIV reported in the literature is variable but may be higher than in the HIV-negative population.

World Health Organization (WHO) and Ugandan national HIV guidelines have recommended the integration of hypertension care into HIV programs since 2014 and 2016, but there has been limited uptake of this recommendation in practice. There have been successful efforts to integrate tuberculosis, malaria, nutrition, maternal-child health, and family planning into HIV programmes in Uganda. In this study, with the goal of identifying opportunities for developing contextually appropriate integrated care models, we mapped the care cascades for both HTN and HIV within a HIV program in Uganda.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above, Having started Antiretroviral therapy between January 2014 and January 2017.

Exclusion Criteria:

* PLHIV receiving treatment from clinics other than the 3 selected sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons Living with HIV (PLHIV) 18 years of age and above who were already diagnosed with HIV and enrolled into HIV care at any of the three sites between January 2014 and January 2017.
Sampling Method: Non-Probability Sample
Enrollment: 1649 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure control | 1 year
  Blood pressure control among Persons living with both HIV and hypertension. Achieving Blood pressure of <140/90mmHg

SECONDARY OUTCOMES:
HIV control | 1 year
  HIV control among persons living with both HIV and hypertension. Defined as HIV Viral suppression. Viral load of <1000 copies/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere University College of Health Sciences, Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months